CLINICAL TRIAL: NCT06468059
Title: Biomechanical Evaluation of a Novel, Compliant Low Profile Prosthetic Foot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Little Room Innovations, LLC (Industry)
Collaborators: Kennesaw State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: R43HD110316 (NIH)
Record Dates: First submitted 2024-06-07; First posted 2024-06-21 (Actual); Results first posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Amputation

STUDY DESIGN:
Who Masked: Participant
Masking Description: The control prosthesis and the experimental prosthesis are covered by a sock to prevent the participant from knowing which has been fit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Layered Low Profile Foot (LPF) vs. Prescribed Ankle (Experimental): In this arm, subjects will first test the LPF and then complete the tests with their prescribed ankle.
  Interventions: Device: Layered Low Profile Foot; Device: Prescribed Ankle
- Prescribed Ankle vs. Layered Low Profile Foot (LPF) (Experimental): In this arm, subjects will first complete the tests with their prescribed ankle and then test the LPF.
  Interventions: Device: Layered Low Profile Foot; Device: Prescribed Ankle

INTERVENTIONS:
Device: Layered Low Profile Foot — The layered LPF is a novel low-profile prosthetic foot that provides compliant behavior while simultaneously exhibiting high mechanical strength.
  Other Names: LPF
Device: Prescribed Ankle — The prescribed ankle is the prosthetic ankle that the subject wears for daily use.
  Other Names: Daily Use Prosthesis

SUMMARY:
The investigators have developed a novel layered low-profile prosthetic foot that is able to provide enhanced compliance without sacrificing strength for individuals with transtibial amputation who have long residual limbs. It is hypothesized that the proposed prosthesis will offer similar benefits to these individuals as comparable higher profile prostheses offer users with shorter residual limbs. The primary goal of this Phase I proposal is to assess the degree to which the proposed prosthesis can provide benefits to prosthesis users in this population, along with characterizing the degree to which the novel prosthesis emulates its taller counterparts.

ELIGIBILITY:
Inclusion Criteria:

1. 18-89 years old
2. unilateral transtibial amputation
3. daily use of a low profile foot
4. cognitive ability to understand and willingness to provide informed consent and follow the study protocol

Exclusion Criteria:

1. unable to perform walking for 2 minutes without an assistive device
2. other health conditions which may prevent them from participating in the study

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-07-16 (Actual); Study Completion 2024-07-16 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Kennesaw State University, Kennesaw, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 subjects were enrolled between 3/21/2024 and 7/16/2024 at Kennesaw State University.
Pre-assignment Details: 6 of 6 patients completed this crossover study.
Period: Overall Study
Arm/Group | Layered Low Profile Foot (LPF) vs. Prescribed Ankle | Prescribed Ankle vs. Layered Low Profile Foot (LPF)
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Layered Low Profile Foot (LPF) vs. Prescribed Ankle | Prescribed Ankle vs. Layered Low Profile Foot (LPF) | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 3 | 2 | 5
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Total Energy Stored (TES)
Description: TES is the amount of energy absorbed by the ankle joint during early and middle stance. It is the integral of the product of joint torque and angular velocity, as determined through inverse dynamics.
Time Frame: through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: Joules
Groups:
- Layered Low Profile Foot (LPF): Layered Low Profile Foot: The layered LPF is a novel low-profile prosthetic foot that provides compliant behavior.
Arm/Group | Prescribed Ankle | Layered Low Profile Foot (LPF)
Number analyzed (Participants) | 6 | 6
Joules | 20.1 (11.2) | 13.3 (6.9)

2. Secondary Outcome: Ankle Quasi-Stiffness (AQS)
Description: AQS is a measure of joint deformation under an applied load. It is extracted from the torque-angle relationship during walking determined through inverse dynamics. The ideal AQS varies from person to person, but in this study we were interested in seeing if the prostheses could achiever lower AQS.
Time Frame: through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: Newton meters per degree
Arm/Group | Prescribed Ankle | Layered Low Profile Foot (LPF)
Number analyzed (Participants) | 6 | 6
Newton meters per degree | 9.8 (2.7) | 9.3 (3.9)

3. Secondary Outcome: Walking Speed
Description: This is the linear rate of change of position when a person walks, typically given in m/s.
Time Frame: through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: Meters per second
Arm/Group | Prescribed Ankle | Layered Low Profile Foot (LPF)
Number analyzed (Participants) | 6 | 6
Meters per second | 1.27 (0.2) | 1.28 (0.2)

4. Secondary Outcome: Likert Scale Rating of Device Satisfaction
Description: A 1 to 10 rating of device satisfaction where the pre-trial perceived device satisfaction of the participant's prescribed ankle is defined as a 5 out of 10. 1 is defined as completely unacceptable, and 10 is defined as ideal performance.
Time Frame: through study completion, an average of 1 day
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Prescribed Ankle | Layered Low Profile Foot (LPF)
Number analyzed (Participants) | 6 | 6
units on a scale | 4.3 (1.5) | 5.2 (1.5)

ADVERSE EVENTS:
Time Frame: For each intervention, the period of time for adverse event monitoring was the 3 to 4 hour period during which the device was worn for the in-lab gait sessions. The participants did not wear the experimental intervention for home or daily use in this study.
Description: The risks associated with study participation are no greater than minimal risk as defined in 45 CFR 46.102(i): "Minimal risk means that the probability and magnitude of harm or discomfort anticipated in the research are not greater in and of themselves than those ordinarily encountered in daily life or during the performance of routine physical or psychological examinations or tests."
Arm/Group | Prescribed Ankle | Layered Low Profile Foot (LPF)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-08-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT06468059/Prot_SAP_ICF_000.pdf